CLINICAL TRIAL: NCT05749549
Title: A Multicenter, Open-Label Phase I/IIa Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics/ Pharmacodynamics and Efficacy of BR1733 Monotherapy in Subjects With Advanced Cancers
Brief Title: Phase I/IIa Study of BR1733 in Subjects With Advanced Cancers
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Blueray Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR1733-101
Record Dates: First submitted 2023-02-16; First posted 2023-03-01 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Advanced Cancer; Follicular Lymphoma; Peripheral T Cell Lymphoma; Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, T-Cell, Peripheral; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BR1733 (Experimental): 25-1200 mg QD or BID
  Interventions: Drug: BR1733

INTERVENTIONS:
Drug: BR1733 — Subjects will receive oral administration of BR1733.

SUMMARY:
This study is a Phase I/IIa, multi-center, open-label study of BR1733 with a dose escalation part followed by a dose expansion part in adult subjects with advanced cancers.

This treatment to characterize the safety, tolerability, PK, PD and preliminary antitumor activity.

The study treatment will be administered until the subject experiences unacceptable toxicity, progressive disease, and/or has treatment discontinued at the discretion of the Investigator or the subject, or due to withdrawal of consent.

DETAILED DESCRIPTION:
This is a multi-center, nonrandomized, open-label study to evaluate the safety, tolerability, pharmacokinetics/ pharmacodynamics, and efficacy of BR1733 in patients with advance cancer, such as recurrent/refractory follicular lymphoma, peripheral T cell lymphoma(PTCL), diffuse large B cell lymphoma(DLBCL) and advance solid tumors.

Phase Ⅰ (Dose Escalation Phase): According to the incidence of DLT in BR1733 tablets in the treatment of advanced cancers, MTD and the Phase 2 clinical trial dose (RP2D) combining PK, PD, efficacy and safety data were determined.

Phase IIa (Dose expansion stage): Evaluate the efficacy and safety of BR1733 monotherapy (Cohorts 1-5) in five separate cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent voluntarily.
2. Subjects with PTCL, DLBCL or advance solid tumors diagnosed by histology or cytology，whose disease progressed after standard treatment or have no standard treatment.
3. ECOG≤2.
4. Expected survival period ≥ 3 months.
5. Adequate organ function reserve at baseline.

Exclusion Criteria:

1. Subjects with symptomatic central nervous system (CNS) metastases or carcinomatous meningitis;
2. Subjects with a history of other primary malignancies within 5 years (except for cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumor), subjects with other primary tumors who had no evidence of disease for 5 years or more and did not require treatment could participate in the study;
3. Subjects with any severe uncontrolled disease such as liver disease such as cirrhosis, decompensated liver disease, kidney failure needs for hemodialysis or peritoneal dialysis, etc.
4. Subjects with HIV disease or a positive HIV test; or active hepatitis.
5. Subjects with organ transplantation (apart from keratoplasty) or allogeneic hematopoietic stem cell transplantation.
6. Subjects with impaired or clinically significant cardiac cerebrovascular disease.
7. Subjects known to be allergic to experimental drugs or similar compounds.
8. Subjects known with psychotropic substance abuse, alcohol or drug abuse, or mental disorders.
9. Any previous treatment with other EED inhibitors (e.g., MAK683, FTX-6058, etc.).
10. Females who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT, Phase Ⅰ only) | 28 day cycle of therapy
  To assess adverse events as dose limiting toxicities as defined by the protocol.
Objective Response Rate (ORR, Phase Ⅱa) | 24 months
  The proportion of patients with a best response of at least partial remission (including partial remission and complete remission) using disease appropriate standardized response criteria.

SECONDARY OUTCOMES:
Halflife (T1/2) of BR1733 monotherapy | 28 day cycle of therapy
  Pharmacokinetics profile of BR1733 (plasma): Halflife (T1/2)
Area under curve (AUC) of BR1733 monotherapy | 28 day cycle of therapy
  Pharmacokinetics profile of BR1733 (plasma): Area under curve (AUC)
Maximum plasma concentration (Cmax) of BR1733 monotherapy | 28 day cycle of therapy
  Pharmacokinetics profile of BR1733 (plasma): Maximum plasma concentration (Cmax)
Area under curve, steady state (AUCss) of BR1733 monotherapy | 28 day cycle of therapy
  Pharmacokinetics profile of continuous medication of BR1733 (plasma): Area under curve, steady state (AUCss)
Maximum plasma concentration, steady state (Cmax,ss) of BR1733 monotherapy | 28 day cycle of therapy
  Pharmacokinetics profile of continuous medication of BR1733 (plasma):
  Maximum plasma concentration, steady state (Cmax,ss)
Clearance/ bioavailability (CL/F) of BR1733 monotherapy | 28 day cycle of therapy
  Pharmacokinetics profile of BR1733 (plasma): Clearance/bioavailability (CL/F)
Incidence and Severity of Adverse Events as a Measure of Safety and Tolerability | Up to 2 years
  Adverse events assessed according to NCI-CTCAE v5.0 criteria.
Duration of Response (DoR) | Up to 2 years
  DoR is defined as the duration (days) from initial response to disease relapse, progression, or death due to any course.
Overall Survival (OS) | Up to 2 years
  OS is defined as the interval of time between the date of first treatment until death, loss to follow up or termination of the study by the sponsor
Progression-free survival (PFS) | Up to 2 years
  PFS is defined as the interval of time between the date of first treatment to the earliest date of disease progression or death which occurs first

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, China